CLINICAL TRIAL: NCT00905268
Title: A Phase III Double-blind, Randomised, Placebo-controlled Study of the Efficacy, Safety and Tolerability of Idebenone in the Treatment of Friedreich's Ataxia Patients
Brief Title: A Study of Efficacy, Safety and Tolerability of Idebenone in the Treatment of Friedreich's Ataxia (FRDA) Patients
Acronym: MICONOS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Santhera Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SNT-III-001
Record Dates: First submitted 2009-05-19; First posted 2009-05-20 (Estimated); Results first posted 2016-06-27 (Estimated); Last update posted 2016-06-27 (Estimated); Status verified 2016-05

CONDITIONS: Friedreich's Ataxia
Keywords: FRDA; idebenone; FRDA disease
MeSH Terms: conditions — Friedreich Ataxia | interventions — idebenone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Group A: Idebenone (Experimental): Patients under/equal 45 kg: idebenone 180 mg/day Patients over 45 kg: idebenone 360 mg/day
  Interventions: Drug: idebenone
- Group B: Idebenone (Experimental): Patients under/equal 45 kg: idebenone 450 mg/day Patients over 45 kg: idebenone 900 mg/day
  Interventions: Drug: idebenone
- C: Idebenone (Experimental): Patients under/equal 45 kg: idebenone 1350 mg/day Patients over 45 kg: idebenone 2250 mg/day
  Interventions: Drug: idebenone
- D: Placebo (Placebo Comparator): placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: idebenone — 12 months of 1 of 3 treatments arms of oral idebenone or placebo.Treatment taken 3 times daily with meals.
  Arms: C: Idebenone; Group A: Idebenone; Group B: Idebenone
Drug: Placebo — 12 months of 1 of 3 treatments arms of oral idebenone or placebo.Treatment taken 3 times daily with meals.
  Arms: D: Placebo

SUMMARY:
The purpose of this trial is to study the efficacy, safety and tolerability of idebenone in 12 months of treatment in children and adults with Friedreich's Ataxia. This is a randomised placebo-controlled double-blind trial conducted in Europe. Efficacy outcomes include measures of neurological impairment and function, and measures of the heart.

DETAILED DESCRIPTION:
Idebenone, a short-chain analogue of Co-enzyme Q10 (CoQ10), has the potential to moderate underlying causes of Friedreich's Ataxia through its antioxidant activity and its role as an electron carrier in the respiratory chain promoting mitochondrial ATP production.

The current 12-month placebo-controlled treatment study in 232 patients aims to confirm the positive effect of idebenone on neurological function, as for instance observed in the recent 48-patient, 6-month NICOSIA study in children, using the International Cooperative Ataxia Rating Scale (ICARS) and the newly developed Friedreich's Ataxia Rating Scale (FARS).

In addition, the study aims to confirm the positive effect on cardiomyopathy associated with FRDA observed in several small studies. Cardiac anatomy and function will be assessed using echocardiography, tissue Doppler imaging and cardiac MRI methods in patients with FRDA cardiomyopathy. In addition exercise capacity, measured as peak workload, will be assessed in patients able to comply with a modified exercise protocol.

ELIGIBILITY:
Inclusion Criteria:

* Documented diagnosis of FRDA with confirmed FRDA mutations
* Patients 8 years of age or older at baseline
* Patients with body weight ≥ 25kg
* Patients who in the opinion of the investigator are able to comply with the requirements of the study, including swallowing the medication
* Negative urine pregnancy test at screening and at baseline (women of childbearing potential)

Exclusion Criteria:

* Treatment with idebenone or Coenzyme Q10 within the past 1 month
* Pregnancy and/or breast-feeding
* Clinically significant abnormalities of clinical haematology or biochemistry including, but not limited to, elevations greater than 1.5 times the upper limit of normal of SGOT, SGPT, or creatinine
* Past or present history of abuse of drugs or alcohol

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 232 (Actual)
Dates: Start 2006-04; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nick Wood, Professor, Principal Investigator — Dept of Molecular Neuroscience, Institute of Neurology. The National Hospital, University college London.
Locations (13):
- Universitätsklinik Innsbruck, Innsbruck, Austria
- Hôpital Erasme - Université Libre de Bruxelles, Brussels, Belgium
- Hôpital de la Salpêtrière - INSERM U679, Neurologie et Thérapeutique expérimentale, Paris, France
- Germany (7):
  - HELIOS Klinikum BerlinBuch, Berlin
  - Neurologische Universitätsklinik und Poliklinik- Universitätsklinikum Bonn, Bonn
  - Klinik II, Neuropädiatrie u.Muskelerkrankungen- Universitätsklinik Freiburg, Freiburg im Breisgau
  - Zentrum für Neurologische Medizin, Göttingen
  - UKE Hamburg Neuropädiatrie-Zentum für Frauen, Kinder und Jugendmedizin, Hamburg
  - Neurologische Klinik- klinikum Grosshadern, München
  - Neurologische Universitätsklinik und Poliklinik, Tübingen
- University Medical Center Groningen, Groningen, Netherlands
- United Kingdom (2):
  - National Hospital for Neurology & Neurosurgery, London
  - University of Newcastle upon Tyne -Mitochondrial Research Group, Newcastle

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group A: Idebenone | Group B: Idebenone | C: Idebenone | D: Placebo
Started | 57 | 57 | 59 | 59
Completed | 53 | 56 | 59 | 57
Not Completed | 4 | 1 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A: Idebenone | Group B: Idebenone | C: Idebenone | D: Placebo | Total
Number analyzed (Participants) | 57 | 57 | 59 | 59 | 232
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.9 (13.7) | 31.6 (13.1) | 30.9 (13.6) | 30.4 (13.3) | 30.9 (13.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 25 | 27 | 32 | 107
  Male | 34 | 32 | 32 | 27 | 125
Region of Enrollment [Number; unit: participants] — The Intent-To-Treat (ITT) population included all randomized subjects who received at least one dose of the study medication and had a confirmed diagnosis of FRDA, did not take idebenone within one month pre-Screening or between Screening and Visit 1, and were not under idebenone treatment at Baseline according to available PK results at Visit 1. The subjects were analyzed as randomized regardless of protocol deviations
  participants
    Germany | 40 | 41 | 39 | 36 | 156
    United Kingdom | 4 | 6 | 6 | 5 | 21
    Austria | 2 | 4 | 2 | 5 | 13
    Belgium | 3 | 1 | 5 | 4 | 13
    France | 5 | 2 | 4 | 6 | 17
    Netherlands | 3 | 3 | 3 | 3 | 12

OUTCOME MEASURES:

1. Primary Outcome: Absolute Change in International Cooperative Ataxia Rating Scale (ICARS) Scores From Baseline Assessment to Week 52
Description: The International Cooperative Ataxia Rating Scale (ICARS) is a commonly used evaluation and is composed of four clinical sub-scores involving the following: posture and gait, limb coordination, speech and oculomotor function.The ICARS score is the total sum of the sub scores and ranges from 0 to 100, with 100 indicative of the most severely affected outcome.
Time Frame: Baseline and week 52
Population: The Intent-To-Treat (ITT) population included all randomized subjects who received at least one dose of the study medication and had a confirmed diagnosis of FRDA, did not take idebenone within one month pre-Screening or between Screening and Visit 1, and were not under idebenone treatment at Baseline according to available PK results at Visit 1.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Group A: Idebenone | Group B: Idebenone | C: Idebenone | D: Placebo
Number analyzed (Participants) | 55 | 55 | 59 | 58
units on a scale | 1.6 (5.85) | 1.7 (6.64) | 1.2 (5.22) | 1.1 (6.76)

2. Secondary Outcome: Absolute Change in Friedreich's Ataxia Rating Scale (FARS) Scores From Baseline Assessment to Week 52
Description: The Friedreich Ataxia Rating Scale (FARS) is made up of a measure of ataxia, and activities of daily living subscale and a neurological subscale. The scores from the three subscales are added to generate a total score ranging from 0 to 159, with a higher score indicating a greater level of disability.
Time Frame: Baseline and week 52
Population: The comparison was carried out in the ITT population, on data imputed using the last observation carried forward (LOCF) method.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Group A: Idebenone | Group B: Idebenone | C: Idebenone | D: Placebo
Number analyzed (Participants) | 54 | 54 | 59 | 58
units on a scale | 0.9 (7.19) | 1.2 (5.24) | 1.4 (5.60) | 0.9 (6.77)

3. Secondary Outcome: Proportion of Patients Improving (Responding) on ICARS by a Clinically Relevant Margin
Description: The International Cooperative Ataxia Rating Scale (ICARS) is a commonly used evaluation and is composed of four clinical sub-scores involving the following: posture and gait, limb coordination, speech and oculomotor function.The ICARS score is the total sum of the sub scores and ranges from 0 to 100, with 100 indicative of the most severely affected outcome.
  ICARS Responder Analysis at Week 52: Percentage of subjects Improving by 2.5 Points or More.
Time Frame: week 52
Population: as for outcome 1
Measure: Number; unit: percentage of patients
Arm/Group | Group A: Idebenone | Group B: Idebenone | C: Idebenone | D: Placebo
Number analyzed (Participants) | 55 | 55 | 59 | 58
percentage of patients | 18.2 | 23.6 | 23.7 | 31

4. Secondary Outcome: Proportion of Patients Improving on Left Ventricular Peak Systolic Strain Rate or Showing a Reduction in Left Ventricular Mass Index (LVMI) With no Worsening in Strain Rate
Description: (In the statistical analysis sub-population presenting with cardiac involvement as defined by the FRDA cardiomyopathy criteria)
Time Frame: 1 year
Population: Subgroup of subjects with cardiac involvement as defined by Friedreich's ataxia cardiomyopathy (FRDA-CM)
Measure: Number; unit: percentage of patients
Arm/Group | Group A: Idebenone | Group B: Idebenone | C: Idebenone | D: Placebo
Number analyzed (Participants) | 36 | 35 | 33 | 34
percentage of patients | 50 | 51.4 | 30.3 | 44.1

5. Secondary Outcome: Change in Peak Systolic Strain Rate From Baseline to Week 52
Description: Mean Change of Peak systolic longitudinal strain rate (PSLSR) from Baseline to Week 52 in subjects with cardiac involvement (FRDA-CM criteria), where positive value in PSLSR is a deterioration and negative value an improvement.
Time Frame: 1 year
Population: Subgroup of subjects with cardiac involvement as defined by Friedreich's ataxia cardiomyopathy (FRDA-CM)
Measure: Mean (Standard Deviation); unit: 1/s
Arm/Group | Group A: Idebenone | Group B: Idebenone | C: Idebenone | D: Placebo
Number analyzed (Participants) | 36 | 35 | 33 | 34
1/s | 0.007 (0.220) | -0.004 (0.265) | 0.085 (0.227) | 0.024 (0.192)

6. Secondary Outcome: Change in Peak Workload From Baseline to Week 52
Description: Assessed by a modified exercise test, in a subset of patients able to undertake this.
  Wpeak has been calculated from the following formula: Workload last fully completed stage + (seconds completed in last stage / 60 * (4 [if arm ergonometry] or 10 [if leg ergonometry])).
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: Watts
Arm/Group | Group A: Idebenone | Group B: Idebenone | C: Idebenone | D: Placebo
Number analyzed (Participants) | 55 | 55 | 59 | 58
Watts | 1.15 (16.362) | -7.41 (34.499) | -6.91 (20.179) | -1.54 (16.509)

ADVERSE EVENTS:
Arm/Group | Group A: Idebenone | Group B: Idebenone | C: Idebenone | D: Placebo
Serious Adverse Events (participants affected / at risk) | 7/57 | 4/57 | 8/59 | 7/59
Other Adverse Events (participants affected / at risk) | 55/57 | 52/57 | 52/59 | 55/59
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A: Idebenone (N=57) | Group B: Idebenone (N=57) | C: Idebenone (N=59) | D: Placebo (N=59)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
diabetes mellitus (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
hypertrophic cardiomyopathy (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
inguinal hernia (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
drug exposure during pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
atrial flutter (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
suparventricular extrasystoles (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
bronchitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
cardiac failure (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
gastrointestinal infection (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
staphylococcal sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
chest pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
suicide attempt (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
influenza like illness (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
procedural pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
renal tubular necrosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
blood creatinine abnormal (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A: Idebenone (N=57) | Group B: Idebenone (N=57) | C: Idebenone (N=59) | D: Placebo (N=59)
palpitations (Cardiac disorders) | 1 (1) | 1 (1) | 3 (3) | 2 (2)
tachycardia (Cardiac disorders) | 3 (3) | 0 (0) | 1 (1) | 2 (2)
vertigo (Ear and labyrinth disorders) | 1 (1) | 2 (2) | 0 (0) | 3 (3)
diarrhea (Gastrointestinal disorders) | 10 (10) | 16 (16) | 10 (10) | 8 (8)
vomiting (Gastrointestinal disorders) | 9 (9) | 5 (5) | 7 (7) | 2 (2)
abdominal pain upper (Gastrointestinal disorders) | 3 (3) | 6 (6) | 6 (6) | 6 (6)
abdominal pain (Gastrointestinal disorders) | 4 (4) | 5 (5) | 2 (2) | 7 (7)
toothache (Gastrointestinal disorders) | 1 (1) | 6 (6) | 4 (4) | 3 (3)
dyspepsia (Gastrointestinal disorders) | 0 (0) | 4 (4) | 1 (1) | 2 (2)
flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
fatigue (General disorders) | 5 (5) | 2 (2) | 2 (2) | 5 (5)
edema peripheral (General disorders) | 0 (0) | 3 (3) | 3 (3) | 1 (1)
pyrexia (General disorders) | 1 (1) | 3 (3) | 0 (0) | 3 (3)
influenza like illness (General disorders) | 1 (1) | 0 (0) | 3 (3) | 0 (0)
nasopharyngitis (Infections and infestations) | 22 (22) | 25 (25) | 21 (21) | 21 (21)
influenza (Infections and infestations) | 7 (7) | 6 (6) | 4 (4) | 5 (5)
bronchitis (Infections and infestations) | 3 (3) | 3 (3) | 4 (4) | 1 (1)
sinusitis (Infections and infestations) | 2 (2) | 1 (1) | 3 (3) | 4 (4)
gastroenteritis (Infections and infestations) | 1 (1) | 2 (2) | 3 (3) | 2 (2)
upper respiratory tract infection (Infections and infestations) | 2 (2) | 1 (1) | 3 (3) | 2 (2)
cystitis (Infections and infestations) | 1 (1) | 4 (4) | 1 (1) | 1 (1)
rhinitis (Infections and infestations) | 2 (2) | 0 (0) | 1 (1) | 3 (3)
fall (Injury, poisoning and procedural complications) | 4 (4) | 7 (7) | 2 (2) | 7 (7)
pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (4) | 7 (7) | 5 (5) | 5 (5)
muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 2 (2) | 5 (5)
headache (Nervous system disorders) | 16 (16) | 20 (20) | 15 (15) | 23 (23)
cough (Respiratory, thoracic and mediastinal disorders) | 11 (11) | 2 (2) | 6 (6) | 6 (6)
oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 6 (6) | 6 (6) | 7 (7)
rash (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1) | 1 (1) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No